CLINICAL TRIAL: NCT04849910
Title: A First-In-Human, Open-Label, Multicenter Study of VOR33 in Patients With Acute Myeloid Leukemia Who Are at High-Risk for Leukemia Relapse Following Hematopoietic Cell Transplantation
Brief Title: Allogeneic Engineered Hematopoietic Stem Cell Transplant (HCT) Lacking the CD33 Protein, and Post-HCT Treatment With Mylotarg, for Patients With CD33+ AML or MDS
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: Vor Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VBP101
Record Dates: First submitted 2021-03-25; First posted 2021-04-19 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-05

CONDITIONS: Leukemia, Myeloid, Acute; Myelodysplastic Syndromes
Keywords: Leukemia; Acute Myeloid Leukemia; AML; Hematopoietic stem cell transplant; HCT; CD33; Allogeneic; Myelodysplastic Syndromes; Myelodysplastic Syndromes with excess blasts; MDS; MDS-EB; Cell therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia | interventions — Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Experimental): VOR33 infusion followed by Mylotarg Dose Level 1
  Interventions: Biological: VOR33; Drug: Mylotarg
- Cohort 2 (Experimental): VOR33 infusion followed by Mylotarg Dose Level 2
  Interventions: Biological: VOR33; Drug: Mylotarg
- Cohort 3 (Experimental): VOR33 infusion followed by Mylotarg Dose Level 3
  Interventions: Biological: VOR33; Drug: Mylotarg

INTERVENTIONS:
Biological: VOR33 — Allogeneic, human leukocyte antigen (HLA) matched, genome edited hematopoietic stem and progenitor cell (HSPC) therapy product lacking the CD33 myeloid protein
Drug: Mylotarg — Infusion of Mylotarg
  Other Names: gemtuzumab ozogamicin

SUMMARY:
This is a Phase 1/2a, multicenter, open-label, first-in-human (FIH) study of VOR33 in participants with AML or MDS who are undergoing human leukocyte antigen (HLA)-matched allogeneic hematopoietic cell transplant (HCT).

DETAILED DESCRIPTION:
High risk acute myeloid leukemia (AML) and myelodysplastic syndromes (MDS) frequently relapses despite hematopoietic stem cell transplant (HCT). Post-HCT targeted therapy to reduce relapse is limited by toxicity to the engrafted cells. VOR33, an allogeneic CRISPR/Cas9 genome-edited hematopoietic stem and progenitor cell (HSPC) therapy product, lacking the CD33 protein, is being investigated for participants with CD33+ AML or MDS at high risk for relapse after HCT to allow post-HCT targeting of residual CD33+ acute AML cells using Mylotarg™ without toxicity to engrafted VOR33 cells. Participants will undergo a myeloablative HCT with matched related or unrelated donor CD34+-selected hematopoietic stem and progenitor cells (HSPCs) engineered to remove CD33 expression (VOR33 product). Mylotarg™ will be given after engraftment for up to 4 cycles. The primary endpoint assessing safety of VOR33 will be the incidence of successful engraftment at 28 days. Part 1 of this study will evaluate the safety of escalating Mylotarg™ dose levels to determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D). Part 2 will expand the number of participants to evaluate the Mylotarg™ RP2D.

ELIGIBILITY:
Inclusion Criteria:

1. Must be ≥18 and ≤70 years of age.
2. Patients with AML must have one of the following groups of features that are known to be a risk factor for leukemia relapse:

   * BM in morphological remission (<5% blasts) with adverse-risk disease related genetics at presentation (according to European Leukemia-Net guidelines [ELN, Döhner 2017]), or
   * Intermediate risk genetics in morphologic remission (<5% blasts) with other recognized high risk criteria such as MRD+ following therapy, or
   * BM with evidence of persistent leukemia 5-10% blasts post induction/salvage therapy. Patients with BM Blast count >10% may participate with Sponsor Medical Monitor approval. (Note: these patients may have disease-related genetics of any risk criteria at presentation), or
   * Any patient in second or greater remission.
3. Patients with MDS must have all of the following:

   * Previous or current IPSS-R score of High or Very High risk; AND
   * Previous or current MDS-IB1 or MDS-IB2 per the 2022 WHO criteria (Khoury 2022)
4. AML sample from the patient must have evidence of CD33 expression (>0%)
5. Candidate for HLA-matched allogeneic HCT using a myeloablative conditioning regimen.
6. Must have a related or unrelated stem cell donor that is a 8/8 match for HLA-A, -B, -C, and -DRB1.
7. Must have adequate performance status and organ function as defined below:

   1. Performance Status: Karnofsky score of ≥70.
   2. Cardiac: left ventricular ejection fraction (LVEF) ≥50%
   3. Pulmonary: diffusing capacity of lung for carbon monoxide (DLCO), forced vital capacity (FVC), and forced expiratory volume in one second (FEV1) ≥66%.
   4. Renal: estimated glomerular filtration rate (GFR) >60 mL/min
   5. Hepatic: total bilirubin <1.5 × ULN, or if ≥1.5 × ULN direct bilirubin <ULN and ALT/AST <1.5 × ULN (per institutional criteria).

Exclusion Criteria:

1. Prior autologous or allogeneic stem cell transplantation.
2. Presence of the following disease-related genetics: t(15; 17)(q22; q21), or t(9; 22)(q34; q11), or other evidence of acute promyelocytic leukemia or chronic myeloid leukemia.
3. Prior treatment with Mylotarg™ (gemtuzumab ozogamicin) in the past 3.5 months.
4. Active central nervous system (CNS) leukemia.
5. Patients diagnosed with Gilbert's syndrome.
6. Uncontrolled bacterial, viral, or fungal infections; or known human immunodeficiency virus (HIV), Hepatitis B, or Hepatitis C infection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Incidence of neutrophil engraftment | Day 28
  Cumulative incidence of patients who achieve neutrophil engraftment (first day of 3 consecutive days of absolute neutrophil count (ANC) ≥500 cells/mm3) by Day 28.

SECONDARY OUTCOMES:
Time to neutrophil engraftment | Up to approximately 28 days
  Time to neutrophil engraftment after HCT from Day 0; calculated as the first day of 3 consecutive laboratory values obtained on separate days where the ANC is ≥500 cells/mm3.
Time to platelet recovery | Up to approximately 60 days
  Time to platelet recovery defined as first day of a sustained platelet count >20,000/ μL with no platelet transfusion in the preceding seven days.
Incidence of acute GVHD Grade (G) G2-G4 and G3-G4 | Up to 24 months
Incidence of chronic GVHD (all and moderate-severe) | Up to 24 months
Incidence of primary and secondary graft failure | Up to 24 months
  Incidence of primary and secondary graft failure measured by day 28 post HCT. Secondary graft failure is defined as initial neutrophil engraftment by Day 28 followed by subsequent decline.
Incidence of toxicities to determine the MTD and RP2D of Mylotarg™ | Approximately day 60 until 24 months
Incidence of transplant-related mortality (TRM) post HCT | Day 100, 12 months, 24 months
Percentage of CD33-negative myeloid cells | Day 28, 60, 100, 180, and Months 12 and 24
  Percent donor myeloid chimerism and CD33-negative myeloid cells in peripheral blood.
Relapse-free Survival (RFS) | Months 12 and 24
  Cumulative incidence of RFS
Overall Survival (OS) | Months 12 and 24
  OS defined as the time from HCT to the date of death from any cause

CONTACTS AND LOCATIONS:
Locations (15):
- United States (14):
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - Stanford Cancer Institute, Stanford, California
  - Miami Cancer Institute, Miami, Florida
  - Winship Cancer Institute Emory University, Atlanta, Georgia
  - The University of Kansas Cancer Center, Fairway, Kansas
  - National Institutes of Health, Clinical Center, Bethesda, Maryland
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine Siteman Cancer Center, St Louis, Missouri
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University Medical Center - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Hôpital Maisonneuve-Rosemont, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Lydeard JR, Lin MI, Ge HG, Halfond A, Wang S, Jones MB, Etchin J, Angelini G, Xavier-Ferrucio J, Lisle J, Salvadore K, Keschner Y, Mager H, Scherer J, Hu J, Mukherjee S, Chakraborty T. Development of a gene edited next-generation hematopoietic cell transplant to enable acute myeloid leukemia treatment by solving off-tumor toxicity. Mol Ther Methods Clin Dev. 2023 Oct 13;31:101135. doi: 10.1016/j.omtm.2023.101135. eCollection 2023 Dec 14. PMID 38027064